CLINICAL TRIAL: NCT04538131
Title: Sensor-Driven Position-Adaptive Spinal Cord Stimulation for Treatment of Gait Disturbance in Parkinson's Disease
Brief Title: Adaptive SCS for Treatment of Gait Disturbance in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Head of Stereotactic and Functional Neurosurgery, Principal Investigator, Clinical Professor, Ruijin Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020 Adaptive SCS PD Gait
Record Dates: First submitted 2020-08-24; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Gait Disorders, Neurologic; Parkinson Disease
MeSH Terms: conditions — Gait Disorders, Neurologic; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- conventional SCS (Active Comparator)
  Interventions: Device: conventional SCS
- sensor-driven position-adaptive SCS (Experimental)
  Interventions: Device: sensor-driven position-adaptive SCS

INTERVENTIONS:
Device: sensor-driven position-adaptive SCS — Medtronic sensor-driven position-adaptive SCS is capable to monitor the position change and change the parameters accordingly, so as to reduce the position change related side effects.
  Arms: sensor-driven position-adaptive SCS
Device: conventional SCS — Conventional SCS can not change the parameter when the body position changes.
  Arms: conventional SCS

SUMMARY:
Spinal cord stimulation (SCS) has been suggested by several research for treating PD gait disturbance. However, the side effects induced by body position change cannot fully addressed by conventional SCS. Medtronic sensor-driven position-adaptive SCS are capable to monitor the position change and change the parameters accordingly, so as to reduce the position change related side effects. Nevertheless, neither the efficacy nor safety of this technique in the treatment of gait disturbance in PD is ever investigated. Therefore, the investigators will conduct a randomized clinical trial to investigate the clinical efficacy and safety of sensor-driven position-adaptive SCS in the treatment of gait disturbance in PD. This study will contribute to find out the safety and efficacy of sensor-driven position-adaptive SCS in the treatment of PD gait disorder, improve patients' quality of life, and reduce the burden on family and society.

DETAILED DESCRIPTION:
The study is a randomized double-blind crossover design aiming to test the short-term efficacy and safety of sensor-driven position-adaptive SCS in the treatment of gait disturbance in patients with PD. More than 1 month after operation, subjects will be randomly assigned into two groups, with one group treated with conventional spinal cord stimulation intervention and the other treated with sensor-driven position-adaptive spinal cord stimulation intervention. Both groups will be followed-up for more than 1 week and receive comprehensive evaluation. A cross-over design will then be applied to eliminate the individual variability until both groups complete another 1 week follow-up. Stimulation parameters and levodopa equivalent daily dose (LEDD) remained during follow-up in both group. Clinical evaluation is assessed by 6-min walk test (6MWT) and timed up-and-go task (TUG) with gait analysis. Quality of life is evaluated by The 5-level EQ-5D. The severity of PIGD is assessed by gait and fall questionnaire (GFQ) , modified fall efficacy scale(MFES), activities-specific balance confidence (ABC) scale and the survey of activities and fear of falling in the elderly (SAFFE ). Within group t test will be made for comparison between two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1,Parkinsonism(including idiopathic Parkinson's disease,Vascular Parkinson's disease, Atypical parkinsonism).
* 2, Aged 45-75 years old, Hoehn & Yahr stage (medication off condition) at 2~4;
* 3, Patients willingly seek surgical treatment for PD gait disturbance；
* 4, Walking disorder with freezing episodes, insufficiently alleviated by oral dopaminergic therapy and/or physiotherapy;
* 5, SCS eligibility has been confirmed by neurologist and neurosurgeon;
* 6, Ability to perform a gait/walking task (under close supervision);
* 7, Informed consent and have good compliance.

Exclusion Criteria:

* 1, Lesion in spinal cord or other surgical contraindications;
* 2, Other neuropsychiatric disorders or relevant medical history; haven't achieved the optimal therapeutic effects of DBS surgery or drug therapy;
* 3, Medical history of stroke, amyotrophic lateral sclerosis or myasthenia gravis; taking prohibited medications (such as lithium, valproate, steroids, adrenergic agonists, etc.);
* 4, Cardiac, renal or other important organs hypofunction or dysfunction, or unstable vital signs;
* 5, Women reporting that they are pregnant;
* 6, Any situation (medical, psychological, social, geographical, etc.) that may endanger patient's life or result in patients withdrawing from the study at present or in the future.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
6-min walk test during the first week (6MWT-1W) | 1 week follow-up
  The 6-min walk test is a test walking over a span of 6 minutes. Gait characters are recorded for further analysis.
timed up-and-go task during the first week (TUG-1W) | 1 week follow-up
  The Timed Up and Go (TUG) test is a performance-based measure of functional mobility that was initially developed to identify mobility and balance impairments in older adults. Gait characters are recorded for further analysis.
6-min walk test during the second week (6MWT-2W) | 2 week follow-up
  The 6-min walk test is a test walking over a span of 6 minutes. Gait characters are recorded for further analysis.
timed up-and-go task during the second week (TUG-2W) | 2 week follow-up
  The 6-min walk test is a test walking over a span of 6 minutes. Gait characters are recorded for further analysis.

SECONDARY OUTCOMES:
EuroQol 5-Dimension, 5-Level Health Scale(EQ-5D-5L) | 1 and 2 week follow-up
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale is a composite of a short descriptive system questionnaire and a visual analogue scale. The EQ-5D-5L descriptive systemmeasures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each state is referred to by a 5-digit code, and the five subscores of the test can be combined to give a summary index value of 0-1, with lower scores representing poorer overall QoLState. The second task component includes a visual analogue scale (VAS) used for rating 'current health state' with a range of 0(worst imaginable health)-100(best imaginable health).
Gait and Fall Questionnaire(GFQ) | 1 and 2 week follow-up
  The FOGQ assesses Freezing of Gait (FOG) severity unrelated to falls in patients with Parkinson's Disease (PD), FOG frequency, disturbances in gait, and relationship to clinical features conceptually associated with gait and motor aspects (e.g., turning).GFQ score has a range of 0 (no gait problems) to 64 (severe gait problems)
Modified Fall Efficacy Scale(MFES) | 1 and 2 week follow-up
  The modified Gait Efficacy Scale (mGES) is a 10-item self-report measure used to assess walking confidence under challenging everyday circumstances.The mFES scale is a visual analog scale in which items are scored from 0 to 10, with 0 meaning "not confident/not sure at all," 5 being "fairly confident/fairly sure," and 10 being "completely confident/completely sure." Total the ratings (possible range = 0 - 140) and divide by 14 to get each subject's mFES score. Scores of < 8 indicate fear of falling, 8 or greater indicate lack of fear.
Activities-specific Balance Confidence (ABC) scale | 1 and 2 week follow-up
  he ABC Scale is a self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness.Items are rated on a 0% to 100% whole number rating scale. Scores of zero represent no confidence; scores of 100 indicate complete confidence. Overall score is calculated by adding item scores and then dividing by the total number of items. Cut-off score of < 69% is predictive of recurrent falls.
Survey of Activities and Fear of Falling in the Elderly (SAFFE ) | 1 and 2 week follow-up
  The Survey of Activities and Fear of Falling in the Elderly (SAFE) was developed to assess these difficulties, and its utility has been demonstrated among the older adults and older people with Parkinson's disease.mSAFFE score has a range of 17-51. Higher scores indicate more fear of failling.

CONTACTS AND LOCATIONS:
Locations (1):
- Functional neurosurgery of Shanghai jiaotong university affiliated Ruijin hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No